CLINICAL TRIAL: NCT02868606
Title: Physiologic Insulin Therapy for the Management of Hyperglycemia in the Hospital
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Donald Brand, PhD, Director of Health Outcomes Research, Winthrop University Hospital
Other Study IDs: 756440-2; R18DK104110 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2016-08-16 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Historical control group (H): Winthrop patients with diabetes hospitalized between August 1, 2010 and March 31, 2011
  Interventions: Other: Sliding-Scale Insulin Therapy
- Intervention group (I): Winthrop patients with diabetes hospitalized between August 1, 2011 and March 31, 2012
  Interventions: Other: Physiologic Insulin Therapy
- Parallel control group (P-sub-H): Patients with diabetes hospitalized between August 1, 2010 and March 31, 2011 at 7 control hospitals located in the New York City metropolitan region
  Interventions: Other: Sliding-Scale Insulin Therapy
- Parallel control group (I-sub-H): Patients with diabetes hospitalized between August 1, 2011 and March 31, 2012 at 7 control hospitals located in the New York City metropolitan region
  Interventions: Other: Sliding-Scale Insulin Therapy

INTERVENTIONS:
Other: Physiologic Insulin Therapy
  Groups: Intervention group (I)
Other: Sliding-Scale Insulin Therapy
  Groups: Historical control group (H); Parallel control group (I-sub-H); Parallel control group (P-sub-H)

SUMMARY:
Many hospitals have begun giving insulin to nearly all patients with diabetes while they are in the hospital even if a patient does not use insulin at home. Controlling blood sugar with insulin when a patient is hospitalized is believed to reduce the risk of complications and death, but research has not demonstrated these benefits except in patients who are critically ill. The purpose of this study, therefore, is to evaluate whether such insulin therapy actually does reduce in-hospital complications, deaths, need for intensive care, or length of stay in the hospital.

DETAILED DESCRIPTION:
The primary aim of the proposed study is to determine if physiologic insulin therapy administered to general hospital inpatients with hyperglycemia favorably affects in-hospital complications and mortality, need for intensive care, or length of stay. The secondary aim is to determine if the magnitude of benefit derived from this therapy differs (a) in patients with known vs. newly diagnosed diabetes, or (b) in medical vs. surgical patients. The study will analyze data from a natural experiment that occurred when the applicant institution introduced universal physiologic insulin therapy as the standard of care for hyperglycemia. A quasi-experimental before-and-after study will compare in-hospital complications, mortality, and resource use in patients with comorbid type 2 diabetes before vs. after implementation of this standard (n≈6400). Outcomes measured at 7 nearby acute-care teaching hospitals during the same two time intervals will provide parallel control data (n≈35,000). Data from the control hospitals will make it possible to evaluate whether temporal changes in patient characteristics or other variables affecting hospitals in the region could explain effects that might otherwise be erroneously attributed to the intervention. Given the high prevalence of comorbid diabetes in the hospital and the possibility that universal physiologic insulin for managing hyperglycemia may not deliver the intended benefit or could even do more harm than good, answering this question is an important goal.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes

Exclusion Criteria:

* Pregnant
* Admitted directly to an intensive care unit
* Length of stay <2 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with type 2 diabetes mellitus admitted to a medical or surgical service
Sampling Method: Probability Sample
Enrollment: 40391 (Actual)
Dates: Start 2015-07; Primary Completion 2017-08-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Transfer to intensive care unit (y/n) | Upon hospital discharge (median length of stay, 5 days)
  Assigned "y" if patient is transferred to an intensive care unit for any length of time; otherwise, assigned "n".

SECONDARY OUTCOMES:
Day-weighted proportion of blood glucose values within target range (100-180 mg/dL) | Upon hospital discharge (median length of stay, 5 days)
Proportion of inpatient days involving any hypoglycemia (blood glucose<70 mg/dL) | Upon hospital discharge (median length of stay, 5 days)
Proportion of inpatient days involving severe hypoglycemia (blood glucose<40 mg/dL) | Upon hospital discharge (median length of stay, 5 days)
Proportion of inpatient days involving any hyperglycemia (blood glucose>200 mg/dL) | Upon hospital discharge (median length of stay, 5 days)
Proportion of inpatient days involving severe hyperglycemia (blood glucose>300 mg/dL) | Upon hospital discharge (median length of stay, 5 days)
Development of any complication (y/n) | Upon hospital discharge (median length of stay, 5 days)
In-hospital death (y/n) | Upon hospital discharge (median length of stay, 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Brand, Ph.D., Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop-University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No